CLINICAL TRIAL: NCT05492786
Title: Alerts With Risk Information to Increase Influenza Vaccinations
Brief Title: High-risk Influenza Vaccine Alert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Massachusetts Institute of Technology (Other); National Institute on Aging (NIA) (NIH); National Bureau of Economic Research, Inc. (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0502; P30AG034532 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Influenza
Keywords: Vaccination; Health Promotion; Health Behavior; Reminder Systems; Economics, Behavioral; Risk Assessment
MeSH Terms: conditions — Influenza, Human; Health Behavior; Behavior | interventions — Caffeine; Risk Factors

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient-participants will not be explicitly told about the different arms, although clinician-participants will see the different arms and may notice these differences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Alert (Active Comparator): Standard flu alert
  Interventions: Behavioral: Alert
- High-risk Alert (Experimental): Flu alert that indicates patient is at high risk for flu and its complications
  Interventions: Behavioral: Alert; Behavioral: Salient alert features; Behavioral: High-risk Text
- High-risk Alert with Risk Factors (Experimental): Flu alert that indicates patient is at high risk for flu and its complications and presents the factors contributing to this high risk
  Interventions: Behavioral: Alert; Behavioral: Salient alert features; Behavioral: High-risk Text; Behavioral: Risk factors

INTERVENTIONS:
Behavioral: Alert — Non-interruptive best practice alert in the electronic health record
Behavioral: Salient alert features — Larger alert header and body font size, use of different font colors and boldface
  Arms: High-risk Alert; High-risk Alert with Risk Factors
Behavioral: High-risk Text — Alert header indicates patient is at high risk for flu and its complications; alert body indicates the percentage of risk (e.g., in the top 3% of risk)
  Arms: High-risk Alert; High-risk Alert with Risk Factors
Behavioral: Risk factors — Alert body indicates the top 3 factors contributing to the high risk
  Arms: High-risk Alert with Risk Factors

SUMMARY:
The purpose of this study is to assess, prospectively, the effect on flu vaccination rates of salient alerts in the electronic health record that indicate a patient's high risk for flu and its complications. The investigators hypothesize that the salient alerts will lead to increased flu vaccination compared with a standard flu alert.

DETAILED DESCRIPTION:
The CDC (Centers for Disease Control) recommends a flu vaccination to everyone aged 6+ months, with rare exception; almost anyone can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death. One barrier to vaccination is a lack of "cues to action," and, in particular, the lack of direct recommendation from medical personnel; this barrier is arguably the most effectively overcome by a simple nudge of clinicians, compared with barriers such as negative attitudes toward vaccination, low perceived utility of vaccination, and less experience with having received the vaccine.

Geisinger partnered with Medial EarlySign (Medial) to develop a machine learning (ML) algorithm to help identify people at risk for serious flu-associated complications based on existing electronic health record data. Eligible at-risk patients will be randomized to an active control group (clinician will be shown a standard flu alert) or one of two experimental groups (clinician will be shown an alert indicating patient's high risk, with or without describing the patient's factors contributing to that risk).

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 18+
* Have been determined to be in the top 20% of risk through Medial's ML algorithm
* Attend an appointment where the flu alert fires (Geisinger sets when flu alerts start and end--between ~9/1/2022 and ~4/30/2023, as well as the trigger conditions for the alert, which includes valid departments and visits and excludes contraindications like Guillain-Barre syndrome)

Clinician Inclusion Criteria:

* Any Geisinger clinician who sees patient-participants in our study for an appointment where their flu shot alert fires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80452 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: https://osf.io/dtkv3/

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinicians: Geisinger clinician who saw patient-participants in our study for an appointment where their flu shot alert fires
Period: Overall Study
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors | Clinicians
Started | 24835 | 24854 | 24912 | 5851
Completed | 24835 | 24854 | 24912 | 5851
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors | Clinicians | Total
Number analyzed (Participants) | 24835 | 24854 | 24912 | 5851 | 80452
Age, Customized [Count of Participants; unit: Participants]
  >=18 and <65 | 15945 | 15783 | 15936 | 5254 | 52918
  >65 | 8890 | 9071 | 8976 | 300 | 27237
  Unknown or not reported | 0 | 0 | 0 | 297 | 297
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 16334 | 16445 | 16368 | 4224 | 53371
  Male | 8501 | 8409 | 8544 | 1322 | 26776
  Unknown or not reported | 0 | 0 | 0 | 305 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1108 | 1201 | 1160 | 165 | 3634
  Not Hispanic or Latino | 23571 | 23503 | 23605 | 5276 | 75955
  Unknown or Not Reported | 156 | 150 | 147 | 410 | 863
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Note: Clinician race/ethnicity data were combined. Clinicians whose race was reported as "Hispanic or Latino" were marked as "Unknown or Not Reported" in the race baseline measure.
  Participants
    Race: American Indian or Alaska Native | 55 | 58 | 60 | 4 | 177
    Race: Asian | 68 | 72 | 83 | 397 | 620
    Race: Native Hawaiian or Other Pacific Islander | 71 | 66 | 93 | 5 | 235
    Race: Black or African American | 871 | 837 | 919 | 129 | 2756
    Race: White | 23613 | 23651 | 23589 | 4686 | 75539
    Race: Two or More | 4 | 5 | 5 | 55 | 69
    Race: Other | 11 | 12 | 15 | 0 | 38
    Race: Unknown or Not Reported | 142 | 153 | 148 | 575 | 1018
Region of Enrollment [Number; unit: participants]
  United States | 24835 | 24854 | 24912 | 5851 | 80452

OUTCOME MEASURES:

1. Primary Outcome: Flu Vaccination
Description: Patient received a flu vaccine (yes/no)
Time Frame: At the 1 day visit
Population: As preregistered, our primary outcome analysis is limited to the first in-person appointment for each patient enrolled in the study. Therefore, this analysis excludes the patients who only attended telehealth appointments during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors
Number analyzed (Participants) | 24257 | 24262 | 24344
Participants | 4459 | 4456 | 4575
Statistical Analysis 1: Comparison: Standard Alert vs High-risk Alert vs High-risk Alert With Risk Factors; Null hypothesis: there is no difference in flu shots for patients whose clinicians were shown alerts with information about their risk status (patients randomized to the High-risk Alert or High-risk Alert with Risk Factors arms) compared with those whose clinicians were shown the standard alert. Alternative hypothesis: patients in the High-risk Alert and High-risk Alert with Risk Factors arms will exhibit improved flu vaccination rates compared with those in the standard Alert arm; Test type: Superiority; p = 0.517, Regression, Linear — The p-value reported is 2-tailed and based on heteroskedasticity-robust standard errors
Statistical Analysis 2: Comparison: High-risk Alert vs High-risk Alert With Risk Factors; Null hypothesis: there is no difference in flu shots for patients whose clinicians were shown alerts the factors that contributed to a patient's high risk (High-risk Alert with Risk Factors arm) compared with those whose clinicians were shown the alert with risk level only (High-risk Alert arm). Alternative hypothesis: patients in the High-risk Alert with Risk Factors arm will exhibit improved flu vaccination rates compared with those in the High-risk Alert arm; Test type: Superiority; p = 0.226, Regression, Linear — The p-value reported is 2-tailed and based on heteroskedasticity-robust standard errors

2. Other Pre Specified Outcome: High Confidence Flu Diagnosis
Description: Patient received a flu diagnosis via a positive polymerase chain reaction [PCR]/antigen/molecular test (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Time Frame: Up to 8 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: "Likely Flu" Diagnosis
Description: Received a "high confidence flu" diagnosis (with positive polymerase chain reaction [PCR]/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test) (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Time Frame: Up to 8 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Flu Complications
Description: Diagnosed with flu-related complications (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Time Frame: Up to 8 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: ER Visits
Description: Number of ER visits from the patient's message appointment date through July 31, 2023
Time Frame: Up to 11 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Hospitalizations
Description: Number of hospitalizations from the patient's message appointment date through July 31, 2023
Time Frame: Up to 11 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: COVID-19 Vaccination Rates
Description: Received at least one COVID-19 vaccination (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Time Frame: Up to 8 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Flu Vaccination During the 2022-2023 Season
Description: Patient receives a flu vaccine (yes/no) during the 2022-23 flu season (from the patient's appointment date through April 30, 2023)
Time Frame: Up to 8 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Flu Vaccination by Sex
Description: Patient received a flu vaccine (yes/no)
Time Frame: At the 1 day visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors
Number analyzed (Participants) | 24257 | 24262 | 24344
Participants
  Female: number analyzed (Participants) | 15928 | 16016 | 15979
  Female | 2817 | 2766 | 2894
  Male: number analyzed (Participants) | 8329 | 8246 | 8365
  Male | 1642 | 1690 | 1681

10. Other Pre Specified Outcome: Flu Vaccination by Race
Description: Patient received a flu vaccine (yes/no)
Time Frame: At the 1 day visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors
Number analyzed (Participants) | 24257 | 24262 | 24344
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 55 | 58 | 60
  American Indian or Alaska Native | 11 | 5 | 9
  Asian: number analyzed (Participants) | 68 | 69 | 82
  Asian | 15 | 20 | 21
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 70 | 66 | 92
  Native Hawaiian or Other Pacific Islander | 10 | 12 | 17
  Black or African American: number analyzed (Participants) | 840 | 810 | 901
  Black or African American | 94 | 90 | 125
  White: number analyzed (Participants) | 23074 | 23093 | 23044
  White | 4302 | 4306 | 4372
  Two or More: number analyzed (Participants) | 4 | 5 | 4
  Two or More | 0 | 1 | 1
  Other: number analyzed (Participants) | 11 | 12 | 15
  Other | 3 | 3 | 4
  Unknown or Not Reported: number analyzed (Participants) | 135 | 149 | 146
  Unknown or Not Reported | 24 | 19 | 26

11. Other Pre Specified Outcome: Flu Vaccination by Ethnicity
Description: Patient received a flu vaccine (yes/no)
Time Frame: At the 1 day visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors
Number analyzed (Participants) | 24257 | 24262 | 24344
Participants
  Hispanic or Latino: number analyzed (Participants) | 1073 | 1178 | 1136
  Hispanic or Latino | 164 | 184 | 172
  Not Hispanic or Latino: number analyzed (Participants) | 23032 | 22939 | 23064
  Not Hispanic or Latino | 4278 | 4244 | 4377
  Unknown or Not Reported: number analyzed (Participants) | 152 | 145 | 144
  Unknown or Not Reported | 17 | 28 | 26

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored. See description.
Description: This is a minimal risk study, and has received expedited IRB review in keeping with 45 CFR § 46.110. EHR and claims data will report inputs (i.e., the subject's assigned arm) and outcomes (i.e., flu vaccination, flu diagnosis, flu-like symptoms). We therefore did not monitor the data for AE/SAEs.
Arm/Group | Standard Alert | High-risk Alert | High-risk Alert With Risk Factors
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT05492786/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT05492786/SAP_000.pdf